CLINICAL TRIAL: NCT00265187
Title: The Prevalence and Clinical Manifestations of Human Metapneumovirus Among Children With Bronchiolitis in Northern Israel.
Brief Title: The Prevalence and Clinical Manifestations of Human Metapneumovirus Among Children With Bronchiolitis.
Status: Completed | Type: Observational
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Dan Miron, MD, HaEmek Medical Center, Afula, Israel
Other Study IDs: 3350105
Record Dates: First submitted 2005-12-13; First posted 2005-12-14 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2006-08

CONDITIONS: Respiratory Tract Infection; Children
Keywords: child, bronchiolitis,
MeSH Terms: conditions — Respiratory Tract Infections; Bronchiolitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Sputum specimens will be obtained from children < 2 years of age and processed by different mode for the HMPV, RSV, Pertussis, Influenza A, B, Parainfluenza 1,2,3, Adenovirus. Clinical and epidemiological data will also be obtained.

DETAILED DESCRIPTION:
The purpose of the study is to asses the various pathogens of bronchiolitis in children and its' clinical manifestations. Prospective study in 3 Medical centers in Northern Israel. Included will be about 200 infants and children < 2 years hospitalized with bronchiolitis. From each child sputum specimen will be obtained and processed for HUMP - PCR, Pertussis - PCR, RSV - ELISA, DFA, PCR, Influenza A, B, Parainfluenza 1,2,3 - DFA, PCR, Adenovirus - DFA. Epidemiological data will be obtained for every child by structured questioner. Clinical data will be daily obtained by scoring system.

ELIGIBILITY:
Inclusion Criteria:Age 0-24 months, hospitalized children, -

Exclusion Criteria:Previous hospitalization, previous RSV immunization, immunocompromised patient, previous inclusion in this study, inclusion in another study.

-

Ages: 1 Day to 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children 0-24 months hospitalized with acute bronchiolitis
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2005-12; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dan Miron, MD, Principal Investigator — HaEmek Medicak Center, Afula, Israel
Locations (3):
- Israel (3):
  - Pediatric department A, HaEmek Medical Center, Afula
  - Maier Hospital, Haifa
  - Pediatric Depart ment , Bnai Zion Hospital, Haifa